CLINICAL TRIAL: NCT06587373
Title: Impact of Traumatic Childbirth on Mother-baby Dyadic Interaction and Maternal Psychological Outcome: a Prospective Study
Acronym: TOPASE+
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: 2024/898
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Parturition Complication
Keywords: MOTHER-BABY DYADIC INTERACTION; MATERNAL PSYCHOLOGICAL MENTAL HEALTH

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — dyadic hair cortisol
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- traumatic childbirth
  Interventions: Other: Assessment of the quality of mother-child dyadic relationships
- non traumatic childbirth
  Interventions: Other: Assessment of the quality of mother-child dyadic relationships

INTERVENTIONS:
Other: Assessment of the quality of mother-child dyadic relationships — Filling out questionnaires

SUMMARY:
While a significant percentage of women in France have difficult pregnancies and negative childbirth experiences, there is still lack of documentation on the impact of these traumatic experiences on maternal health and mother-child relationships. Few studies have focused on the mental health of mothers, despite traumatic experiences being a risk factor for post-traumatic stress, depressive disorders, and suicide. The findings also highlights the maternal withdrawals and intrusions in interaction with the child, which are associated with guilt and feelings of helplessness, a risk to the emotional regulation of the child. Additionally, avoidance symptoms resulting from traumatic experiences delay mothers' seeking help and the early management of dysfunctional interactions. Therefore, assessing the mother-child interactions is important in understanding perinatal psychopathology.

DETAILED DESCRIPTION:
The population include the mother-infant dyads participated in the previous study TOPASE).

The study population comprises 2 groups: a group of women who have experienced a traumatic birth and/or a birth perceived as traumatic by the midwives, and a group of women who have experienced a non-traumatic birth and/or a birth perceived as non-traumatic by the midwives.

The aim of this study is to analyze the impact of traumatic childbirth on the quality of mother-baby dyadic interaction and describe the impact of traumatic childbirth on the mother's mental health and the child's psychomotor and social-emotional development.

ELIGIBILITY:
Concerning the mother :

Inclusion Criteria:

* Women who participated in the TOPASE study
* Non-opposition indicating that the subject agrees to participate in the study and to abide by the requirements and restrictions inherent to this study (including hair sampling for mother and child)
* Affiliation with a French social security scheme or beneficiary of such a scheme
* Women belonging to the "Traumatic delivery" group: QEVA and/or QETRAS score less than or equal to the first quartile
* Women belonging to the "Non-traumatic delivery" group: QEVA and/or QETRAS score greater than or equal to the third quartile

Exclusion Criteria:

* Persons deprived of their liberty by a judicial or administrative decision; persons under compulsory psychiatric care; persons admitted to a health or social establishment for purposes other than research.
* adults under legal protection or unable to express their consent
* Subjects in the exclusion period of another study or in the "national volunteer file".
* Subject unlikely to cooperate with the study and/or poor cooperation anticipated by the investigator
* Refusal to take hair samples from the dyad
* Refusal of video recording of dyad
* Language barrier preventing understanding of instructions
* Cognitive impairment preventing understanding of study instructions
* Women whose child had been hospitalized in intensive care for more than a week or had died

Concerning the child :

Inclusion Criteria:

* No opposition from holders of parental authority

Exclusion Criteria:

* Child with organic malformation and/or objectified genetic anomaly

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women from the TOPASE study, having obtained a QEVA and/or QETRAS score either ≤ the first quartile (traumatic childbirth group) or ≥ the third quartile (non-traumatic childbirth group) will be contacted in random order (a random draw using R software until the desired number of women is obtained) at 15 months (+/-3 months) after delivery by a midwife from the gynecology-obstetrics department in order to propose participation in the study
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-01-02 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Quality of mother-baby dyadic interactions assessed by Coding Interactive Behavior | 15 months (+/- 3 months) postpartum
  Assessed by Coding Interactive Behavior subscores:
  * dyadic reciprocity
  * mother-infant avoidance
  * mother and child engagement
  The rating grid includes 43 items: 22 for the adult, 16 for the child and 5 for the dyad.
  The rating is carried out after observing the entire sequence and reflects the observer's judgment taking into account the relative levels of specific behaviors, the nature of affective/attentional states, reciprocity and adaptation of partners in the interaction between them.
  For each item, the clinician assigns a score between 1 and 5 (level 1 being a low occurrence of a behavior or emotion and 5 a high level of appearance of the characteristic of the element in the interaction).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Besançon, Besançon, France

REFERENCES:
- [Background] Ayers, S., Eagle, A., & Waring, H. (2006). The effects of childbirth-related post-traumatic stress disorder on women and their relationships: A qualitative study. Psychology, Health & Medicine, 11(4), 389-398. https://doi.org/10.1080/13548500600708409 Ayers, S., Joseph, S., McKenzie-McHarg, K., Slade, P., & Wijma, K. (2008). Post-traumatic stress disorder following childbirth: Current issues and recommendations for future research. Journal of Psychosomatic Obstetrics and Gynaecology, 29(4), 240-250. https://doi.org/10.1080/01674820802034631 Berger, M., Castellani, C., Ninoreille, K., Basset, T., Frere-Meusnier, D., & Rigaud, C. (2010). Stress dus aux traumatismes relationnels précoces: Conséquences cérébrales de la perturbation de la sécrétion du cortisol sanguin chez les nourrissons. Neuropsychologie, 58(5), 282-292. https://doi.org/10.1016/j.neurenf.2009.09.003 Brockington, I. F., Oates, J., George, S., Turner, D., Vostanis, P., Sullivan, M., Loh, C., & Murdoch, C. (2001). A Screening Questionnaire for mother-infant bonding disorders. Archives of Women's Mental Health, 3(4), 133-140. https://doi.org/10.1007/s007370170010 Chabbert, M., & Wendland, J. (2016). Le vécu de l'accouchement et le sentiment de contrôle perçu par la femme lors du travail: Un impact sur les relations précoces mère-bébé ? Revue de Médecine Périnatale, 8(4), 199-206. https://doi.org/10.1007/s12611-016-0380-x Chasson, M., & Taubman - Ben-Ari, O. (2023). The Maternal Disintegrative Responses Scale (MDRS): Development and initial validation. Journal of Clinical Psychology, 79(2), 415-430. https://doi.org/10.1002/jclp.23414 Cox, J. L., Chapman, G., Murray, D., & Jones, P. (1996). Validation of the Edinburgh Postnatal Depression Scale (EPDS) in non-postnatal women. Journal of Affective Disorders, 39(3), 185-189. Cox, J. L., Murray, D., & Chapman, G. (1993). A Controlled Study of the Onset, Duration and Prevalence of Postnatal Depression. British Journal of Psychiatry, 163(1), 27-31. https://doi.org/10.1192/bjp.163.1.27 Davies, J., Slade, P., Wright, I., & Stewart, P. (2008). Posttraumatic stress symptoms following childbirth and mothers' perceptions of their infants. Infant Mental Health Journal, 29(6), 537-554. https://doi.org/10.1002/imhj.20197 Dekel, S., Ein-Dor, T., Dishy, G. A., & Mayopoulos, P. A. (2020). Beyond postpartum depression: Posttraumatic stress-depressive response following childbirth. Archives of Women's Mental Health, 23(4), 557-564. https://doi.org/10.1007/s00737-019-01006-x Dekel, S., Stuebe, C., & Dishy, G. (2017). Childbirth Induced Posttraumatic Stress Syndrome: A Systematic Review of Prevalence and Risk Factors. Frontiers in Psychology, 8, 560. https://doi.org/10.3389/fpsyg.2017.00560 Diagnostic and statistical manual of mental disorders: DSM-5TM, 5th ed. (pp. xliv, 947). (2013). American Psychiatric Publishing, Inc. https://doi.org/10.1176/appi.books.9780890425596 Ertan, D., Hingray, C., Burlacu, E., Sterlé, A., & El-Hage, W. (2021). Post-traumatic stress disorder following childbirth. BMC Psychiatry, 21(1), 155. https://doi.org/10.1186/s12888-021-03158-6 Feldman, R. (1998). Coding interactive behavior manual. Unpublished Manual. Ferber, S. G., Feldman, R., Kohelet, D., Kuint, J., Dollberg, S., Arbel, E., & Weller, A. (2005). Massage therapy facilitates mother-infant interaction in premature infants. Infant Behavior and Development, 28(1), 74-81. https://doi.org/10.1016/j.infbeh.2004.07.004 Fournier, A., & Bérubé, A. (2018). La qualité de l'interaction mère-enfant et le rôle du cortisol: Portrait d'une population vivant en contexte de vulnérabilité. Frankham, L. J., Thorsteinsson, E. B., & Bartik, W. (2023). Birth related PTSD and its association with the mother-infant relationship: A meta-analysis. Sexual & Reproductive Healthcare, 38, 100920. https://doi.org/10.1016/j.srhc.2023.100920 Garthus-Niegel, S., Horsch, A., Handtke, E., von Soest, T., Ayers, S., Weidner, K., & Eberhard-Gran, M. (2018). The Impact of Postpartum Posttraumatic Stress and Depression Symptoms on Couples' Relationship Satisfaction: A Population-Based Prospective Study. Frontiers in Psychology, 9, 1728. https://doi.org/10.3389/fpsyg.2018.01728 Guedeney, A., & Tereno, S. (2012). La vidéo dans l'observation d'évaluation et d'intervention en santé mentale du jeune enfant: Un outil pour la transmission. Transmission - Strasbourg 2010 - Seconde Partie, 60(4), 261-266. https://doi.org/10.1016/j.neurenf.2011.12.001